CLINICAL TRIAL: NCT00516126
Title: Goal-orientated Therapy of Perioperative Disturbance in Hemostasis With MULTIPLATE and ROTEM in Cardiac Surgery Patients Under Platelets Inhibitors
Brief Title: Goal-orientated Therapy of Perioperative Disturbance in Hemostasis in Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Daniel Bolliger, PD Dr. Daniel Bolliger, University Hospital, Basel, Switzerland
Other Study IDs: 194/06
Record Dates: First submitted 2007-08-13; First posted 2007-08-14 (Estimated); Last update posted 2013-01-11 (Estimated); Status verified 2013-01

CONDITIONS: Coronary Artery Bypass Graft Triple Vessel; Blood Coagulation Disorders
Keywords: hemostasis monitoring; perioperative blood loss
MeSH Terms: conditions — Blood Coagulation Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Point-of-Care managed: This arm includes all patients in which the hemostatic therapy is guided by POC devices e.g. MULTIPLATE (a platelet function analyzer) or ROTEM (thromboelastometry)
- Conventional hemostasis lab managed: This arm includes all patients in which the hemostatic therapy is guided by conventional hemostasis laboratory data e.g. INR, aPTT, fibrinogen concentration, platelet count but no POC devices e.g. MULTIPLATE (a platelet function analyzer) or ROTEM (thromboelastometry)

SUMMARY:
Aim of this study is to investigate whether patients preoperatively treated with acetylsalicylic acid and/or clopidogrel have fewer perioperative bleeding and lower amounts of blood substitution when managed by ROTEM (whole blood coagulation analyzer) and MULTIPLATE (thrombocyte function analyzer).

ELIGIBILITY:
Inclusion Criteria:

* written consent

Exclusion Criteria:

* no written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2009-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Perioperative blood loss | 24 hours

SECONDARY OUTCOMES:
perioperative substitution with erythrocyte concentrates, thrombocyte concentrates or fresh frozen plasma | 24 hours and 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Miodrag Filipovic, PhD, MD, Study Director — Department of Anesthesia, University Hospital Basel, CH-4031 Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, CH, Switzerland